CLINICAL TRIAL: NCT00445445
Title: Longitudinal Changes in Mammographic Density and Risk of Breast Cancer
Brief Title: Changes in Breast Density and Breast Cancer Risk in Women With Breast Cancer and in Healthy Women
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE1105; P30CA043703 (NIH); CASE1105 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Time perspective: Prospective and retrospective. Blood and urine samples will be processed in our lab and stored in a -80 degree freezer until needed. Urine samples will be assessed for levels of bisphenol-A and remaining samples of urine and blood will be stored for future projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Histologically confirmed breast cancer that was diagnosed between the years 2002-2004
  Interventions: Other: physiologic testing; Other: screening questionnaire administration; Procedure: breast imaging study; Procedure: radiomammography; Procedure: study of high risk factors
- Healthy participants: Healthy participant who is receiving routine medical care (e.g., screening mammograms. Healthy participants are frequency-matched by age (± 2 years) and ethnicity.
  Interventions: Other: physiologic testing; Other: screening questionnaire administration; Procedure: breast imaging study; Procedure: radiomammography; Procedure: study of high risk factors

INTERVENTIONS:
Other: physiologic testing — Urine samples will be assessed for levels of bisphenol-A
Other: screening questionnaire administration — Patients and healthy participants complete a self-administered questionnaire providing detailed information on breast cancer risk factors, including demographics, behavioral and lifestyle factors, reproductive history, family history of breast cancer, comorbidities, medication and hormone replacement therapy use, and breast cancer screening history. This information is then cross-validated with documented data abstracted from medical records to provide a longitudinal and historical framework for assessing individual risk.
Procedure: breast imaging study — Mammographic density (MD) assessment: Patients and healthy participants are evaluated for patterns of longitudinal change in MD and subsequent breast cancer risk by retrospective review of screening mammograms performed prior to breast cancer diagnosis.
Procedure: radiomammography — Mammographic density (MD) assessment: Patients and healthy participants are evaluated for patterns of longitudinal change in MD and subsequent breast cancer risk by retrospective review of screening mammograms performed prior to breast cancer diagnosis.
Procedure: study of high risk factors — * Questionnaire: Patients and healthy participants complete a self-administered questionnaire providing detailed information on breast cancer risk factors, including demographics, behavioral and lifestyle factors, reproductive history, family history of breast cancer, comorbidities, medication and hormone replacement therapy use, and breast cancer screening history. This information is then cross-validated with documented data abstracted from medical records to provide a longitudinal and historical framework for assessing individual risk.
  * Mammographic density (MD) assessment: Patients and healthy participants are evaluated for patterns of longitudinal change in MD and subsequent breast cancer risk by retrospective review of screening mammograms performed prior to breast cancer diagnosis.

SUMMARY:
RATIONALE: Studying mammograms for breast density changes over time may help doctors predict breast cancer risk.

PURPOSE: This natural history study is looking at changes in breast density and gathering health information over time to assess breast cancer risk in women with breast cancer and in healthy women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize each woman's individual mammographic density (MD) longitudinal change trajectory in women with breast cancer and in healthy female participants to assess within-individual MD longitudinal change and breast cancer risk.
* Examine whether these patients or healthy participants manifest different patterns of within-individual change in MD and evaluate predictors of across-individual differences.
* Determine whether the developmental profile of MD differs systematically between these patients and healthy participants.

OUTLINE: This is a prospective, retrospective, controlled study. Patients and healthy participants are frequency-matched by age (± 2 years) and ethnicity.

* Questionnaire: Patients and healthy participants complete a self-administered questionnaire providing detailed information on breast cancer risk factors, including demographics, behavioral and lifestyle factors, reproductive history, family history of breast cancer, comorbidities, medication and hormone replacement therapy use, and breast cancer screening history. This information is then cross-validated with documented data abstracted from medical records to provide a longitudinal and historical framework for assessing individual risk.
* Mammographic density (MD) assessment: Patients and healthy participants are evaluated for patterns of longitudinal change in MD and subsequent breast cancer risk by retrospective review of screening mammograms performed prior to breast cancer diagnosis.

PROJECTED ACCRUAL: A total of 1500 patients and 1500 healthy participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the University Hospitals Breast Center and primary care clinics within the University Hospitals system
* Have at least 3 screening mammograms since 1994
* for cases, diagnosis with breast cancer between 2004-2006

Exclusion criteria:

* having had irregular screening (less than 3 mammorgrams since 1994)
* Having breast implants
* Known carriers of BRCA1/BRCA2 genes
* Unable to give written consent

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer cases diagnosed after 1994 and equal number of frequency-matched (by age within 2 years and ethnicity) controls. Cases and eligible controls with at least 3 screening mammograms since 1994 will be recruited through the University Hospitals Breast Center, and primary care clinics within the University Hospitals Health System (UHHS). The restriction of 3 or more screening mammograms will allow us to adequately model the longitudinal change patterns.
Sampling Method: Probability Sample
Enrollment: 2201 (Actual)
Dates: Start 2007-01-10 (Actual); Primary Completion 2014-07-21 (Actual); Study Completion 2014-07-21 (Actual)

PRIMARY OUTCOMES:
Within-individual mammographic density (MD) longitudinal change and breast cancer risk | cancer cases diagnosed within the last 3 years (2004-2006).
Patterns of within-individual longitudinal change in MD | cancer cases diagnosed within the last 3 years (2004-2006)
Predictors of across-individual differences in MD change | cancer cases diagnosed within the last 3 years (2004-2006)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Thompson, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (8):
- United States (8):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Monarch, Mayfield Heights, Ohio
  - UH-LUICC, Mentor, Ohio
  - UH-Southwest, Middleburg Heights, Ohio
  - UH-Chagrin Highlands Orange Village Ohio 44122, Orange, Ohio
  - UH-Firelands, Sandusky, Ohio
  - UH-Green Road, South Euclid, Ohio
  - UH-Westlake, Westlake, Ohio